CLINICAL TRIAL: NCT05683964
Title: Understanding the Interaction Between Androgen Receptor Signaling and Prostate-Specific Membrane Antigen Expression
Brief Title: Androgen Receptor Signaling and Prostate-Specific Membrane Antigen Expression
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, David J. Einstein, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-441
Record Dates: First submitted 2022-12-19; First posted 2023-01-13 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Prostate Adenocarcinoma; Prostate Cancer; Metastatic Hormone-Sensitive Prostate Cancer (mHSPC)
Keywords: Prostate Adenocarcinoma; Prostate Cancer; Metastatic Hormone-Sensitive Prostate Cancer (mHSPC)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; darolutamide; enzalutamide; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Androgen Receptor Antagonist Monotherapy (Experimental): * Participants will receive pre-determined doses of apalutamide, darolutamide, or enzalutamide per standard care.
  * Participants will undergo Prostate-Specific Membrane Antigen (PSMA) PET/CT scans at weeks 1 and 4.
  Interventions: Drug: Apalutamide [Erleada], darolutamide [Nubeqa], or enzalutamide [Xtandi]; Diagnostic Test: Prostate-Specific Membrane Antigen (PSMA) PET/CT Scan

INTERVENTIONS:
Drug: Apalutamide [Erleada], darolutamide [Nubeqa], or enzalutamide [Xtandi] — per standard care
Diagnostic Test: Prostate-Specific Membrane Antigen (PSMA) PET/CT Scan — Per standard care

SUMMARY:
The goal of this research study is to determine whether hormonal therapies used early in the course of prostate cancer could increase the amount of Prostate-Specific Membrane Antigen (PSMA) as detected by PET/CT scans for participants with recurrent prostate cancer. This study will measure PSMA levels using standard PET/CT scans and participants will receive standard-of-care androgen receptor antagonist monotherapy.

The names of the treatment interventions involved in this study are:

* Androgen receptor antagonist monotherapy.
* PSMA PET/CT scan

It is expected that about 15 people will take part in this research study.

Participation in this research study is expected to last about 4 weeks.

DETAILED DESCRIPTION:
This research study is a pilot study, and it is the first time investigators are directly examining the effect of standard androgen receptor antagonists on Prostate-Specific Membrane Antigen (PSMA) expression for participants with recurrent, asymptomatic, metastatic hormone-sensitive prostate cancer (mHSPC). This study will measure PSMA levels using standard PET/CT scans and participants will receive standard-of-care androgen receptor antagonist monotherapy.

The research study procedures include screening for eligibility, study imaging and evaluations, blood collections, and follow up visits.

The names of the treatment interventions involved in this study are:

* Androgen receptor antagonist monotherapy.
* PSMA PET/CT scan

The U.S. Food and Drug Administration (FDA) has approved apalutamide, darolutamide, and enzalutamide for the treatment of prostate cancer.

It is expected that about 15 people will take part in this research study.

Participation in this research study is expected to last about 4 weeks.

Funding for this research study is provided by a philanthropic gift.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 40 or higher with prostate cancer that has been previously treated with primary definitive local therapies (prostatectomy with or without salvage radiation, or primary prostate radiation) and subsequently experiencing rising PSA meeting criteria for biochemical failure (PSA >0.2 ng/dL x2 following prostatectomy, or PSA > 2 + nadir value following primary radiation).
* PSMA PET/CT (Ga68, piflutolastat F-18, or other FDA-approved tracer) during time of biochemical recurrence, and within 6 weeks of registration, showing at least one lesion suspicious for recurrent prostate cancer based on size and/or SUV.
* Testosterone >100 ng/dL within 6 months prior to enrollment with no intervening hormonal therapies.
* Assigned by treating physician to receive standard-of-care AR antagonist monotherapy, using FDA-approved apalutamide, darolutamide, or enzalutamide.

Exclusion Criteria:

* High disease burden, significant symptoms of disease, or other clinical situation requiring medical/surgical castration and/or docetaxel during the time of the study.
* Not suitable for AR antagonist therapy (e.g. inability to swallow pills, poor adherence, advanced liver disease, prohibitive co-payment without available patient assistance funding, contraindicated drug-drug interaction).
* Older-generation AR antagonists (e.g. bicalutamide) are not allowed on study.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 15 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with New Lesions (Flare) | week 1
  Defined as the percentage of patients having the appearance of at least one new suspicious lesion or increase in SUV max relative to each individual's baseline.
Proportion of Participants with New Lesions (Flare) | week 4
  Defined as the percentage of patients having the appearance of at least one new suspicious lesion or increase in SUV max relative to each individual's baseline.

SECONDARY OUTCOMES:
Changes in tumor size | week 1
  Defined as maximum diameter of lesions for up to 5 target lesions. Standardized Uptake Value Max and Mean.
Changes in tumor size | week 4
  Defined as maximum diameter of lesions for up to 5 target lesions. Standardized Uptake Value Max and Mean.
Changes in tumor SUV | week 1
  For up to 5 target lesions. Standardized Uptake Value Max and Mean.
Changes in tumor SUV | week 4
  For up to 5 target lesions. Standardized Uptake Value Max and Mean.
Changes in serum PSA | week 1
Changes in serum PSA | week 4

CONTACTS AND LOCATIONS:
Overall Officials: David Einstein, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu